CLINICAL TRIAL: NCT00723333
Title: Chart Review of Reduced Intensity Conditioning (RIC) Allogeneic Transplants in Elderly Patients With Myelofibrosis.
Brief Title: Bone Marrow Transplant Chart Review for RIC
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Collaborators: Fred Hutchinson Cancer Center (Other); Baylor College of Medicine (Other); M.D. Anderson Cancer Center (Other)
Responsible Party: Josef T. Prchal, MD, University of Utah
Other Study IDs: 29021
Record Dates: First submitted 2008-07-24; First posted 2008-07-28 (Estimated); Last update posted 2009-10-12 (Estimated); Status verified 2009-10

CONDITIONS: Myelofibrosis
Keywords: Bone Marrow Transplant; Myelofibrosis; Stem Cell Transplant; Allogenic Transplant
MeSH Terms: conditions — Primary Myelofibrosis | interventions — Bone Marrow Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Affected Group: Patients > 60 years of age with Primary Myelofibrosis that have undergone an allogeneic transplant
  Interventions: Procedure: Reduced Intensity Conditioning (RIC) Allogenic Transplant

INTERVENTIONS:
Procedure: Reduced Intensity Conditioning (RIC) Allogenic Transplant — Reduced Intensity Conditioning (RIC) Regimen Allogenic Stem Cell Transplant
  Other Names: Stem Cell Transplants; Bone Marrow Transplants; Mini Transplants

SUMMARY:
We will evaluate the records of 30 patients that have undergone allogeneic transplant, specifically looking at engraftment rate, relapse rate, disease free survival, overall survival, causes of death and other pertinent statistics. We will compare the outcomes to appropriate historical controls.

DETAILED DESCRIPTION:
Primary myelofibrosis (PMF) is among the Philadelphia Chromosome Negative Myeloproliferative Disorders. This diagnosis can be present at a patient's initial diagnosis or it can arise out of preceding Polycythemia Vera or Essential Thrombocythemia. While the clinical course is variable, it is defined by varying degrees of splenomegaly, anemia, fatigue and other constitutional symptoms. Patients with PMF are at increased risk of acute leukemia, bone marrow failure and thrombosis. Currently, the only curative treatment for PMF is allogeneic stem cell transplant. However, as the median age at diagnosis is in the mid to late 60s, most patients are no longer candidates for transplant due to their age and/or other comorbid illnesses.

Unfortunately, all other treatments for PMF are palliative in nature and often of limited efficacy. Over the last several years, many advances have occurred that have increased the safety and improved the outcomes of allogeneic transplants. Perhaps most important has been the ongoing refinement of reduced intensity conditioning (RIC) regimens prior to transplant. Over the last few years, many groups have published data suggesting that these RIC transplants can be very effective in the treatment of PMF and it is felt to be a potentially curative procedure. However, the vast majority of these data are reported in persons younger than 65 years old. The current protocol for RIC transplant for PMF available at the University of Utah excludes patients older than the age of 65.

We would like to see if there is sufficient successful experience with transplant in persons older than 60 years old (including many older than 65 years of age) to justify the creation of a clinical trial using RIC regimens in this older age group. We will be reviewing the medical records of approximately 30 patients at four different institutions:

* University of Utah/Huntsman Cancer Hospital
* Fred Hutchinson Cancer Research Center
* Baylor College of Medicine
* M.D. Anderson Cancer Centers

We will evaluate: engraftment rate, relapse rate, disease free survival, overall survival, causes of death and other pertinent statistics. We will compare the outcomes to appropriate historical controls. We hypothesize that RIC regimens may be justifiably safe in older patients with PMF and hope that our data will allow the development of a corollary clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* > 60 years of age
* Diagnosed with Primary Myelofibrosis
* Undergone Allogeneic Transplant

Exclusion Criteria:

* Any subjects not meeting the criteria above

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients > 60 years of age with Primary Myelofibrosis that have undergone an allogeneic transplant
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2008-05; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Evaluation of engraftment rate, relapse rate, disease free survival, overall survival, causes of death and other pertinent statistics. Data will be compared to appropriate historical controls. | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Josef T Prchal, MD, Principal Investigator — University of Utah
Locations (4):
- United States (4):
  - Baylor College of Medicine, Houston, Texas
  - M.D. Anderson Cancer Centers, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - Fred Hutchinson Cancer Research Center, Seattle, Washington

REFERENCES:
- [Background] Hoffman R, Rondelli D. Biology and treatment of primary myelofibrosis. Hematology Am Soc Hematol Educ Program. 2007:346-54. doi: 10.1182/asheducation-2007.1.346. PMID 18024650
- [Background] Mesa RA, Silverstein MN, Jacobsen SJ, Wollan PC, Tefferi A. Population-based incidence and survival figures in essential thrombocythemia and agnogenic myeloid metaplasia: an Olmsted County Study, 1976-1995. Am J Hematol. 1999 May;61(1):10-5. doi: 10.1002/(sici)1096-8652(199905)61:13.0.co;2-i. PMID 10331505
- [Background] Rondelli D, Barosi G, Bacigalupo A, Prchal JT, Popat U, Alessandrino EP, Spivak JL, Smith BD, Klingemann HG, Fruchtman S, Hoffman R; Myeloproliferative Diseases-Research Consortium. Allogeneic hematopoietic stem-cell transplantation with reduced-intensity conditioning in intermediate- or high-risk patients with myelofibrosis with myeloid metaplasia. Blood. 2005 May 15;105(10):4115-9. doi: 10.1182/blood-2004-11-4299. Epub 2005 Jan 25. PMID 15671439